CLINICAL TRIAL: NCT06226103
Title: Effectiveness Of Computer-Based Cognitive Training Combined With Aerobic Training in Age-Related Cognitive Decline
Brief Title: Effectiveness Of Computer-Based Cognitive Training in Age-Related Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Dr. Mohammad Abu Shaphe, Associate Professor, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC-45/06/919
Record Dates: First submitted 2024-01-05; First posted 2024-01-26 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Age-related Cognitive Decline
Keywords: Cognition; Computer Based Cognitive Training; Aerobic Training; Exercises
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Group (Aerobic Exercise and Computerized Cognitive Training) (Experimental): Aerobic Exercise (AE) included walk briskly, increasing intensity and duration progressively. The first week they had to walk 30 min per day, 3 days per week, up to 9-10 on the Borg Rating of Perceived Exertion Scale (BRPES; Borg, 1982) perceived as light intensity; during the second week, the duration was increased to 45 min and the intensity 9-10 and frequency (3 days per week) were maintained; the following 10 weeks they maintained the duration (45 min) and frequency (3 days per week) and increased the intensity up to 12-14 on BRPES perceived as moderate-high effort.
  Computerized Cognitive Training (CCT) included a multidomain computer-based cognitive training using the brainHQ software in sessions of 45 min, 3 days per week for 12 weeks. Cognitive tasks targeted attention, recognition, colour and shape, identification, calculation, visual perception, visual spatial processing, memory, and executive function).
  Interventions: Other: Aerobic Exercise and Computerized Cognitive Training
- Control Group (Active Comparator): Participants were exposed to balancing, coordination, stretching, and core exercises. Additionally, they attended brain health lectures to provide a comparative non-interactive cognitive engagement. Both the exercises and lectures were scheduled similar to the intervention group over 12 weeks.
  Interventions: Other: Conventional Exercises and Brain health lectures

INTERVENTIONS:
Other: Aerobic Exercise and Computerized Cognitive Training — Aerobic Exercise (AE) included walk briskly, increasing intensity and duration progressively. The first week they had to walk 30 min per day, 3 days per week, up to 9-10 on the Borg Rating of Perceived Exertion Scale (BRPES; Borg, 1982) perceived as light intensity; during the second week, the duration was increased to 45 min and the intensity 9-10 and frequency (3 days per week) were maintained; the following 10 weeks they maintained the duration (45 min) and frequency (3 days per week) and increased the intensity up to 12-14 on BRPES perceived as moderate-high effort.
  Computerized Cognitive Training (CCT) included a multidomain computer-based cognitive training using the brainHQ software in sessions of 45 min, 3 days per week for 12 weeks. Cognitive tasks targeted attention, recognition, colour and shape, identification, calculation, visual perception, visual spatial processing, memory, and executive function.
  Arms: Interventional Group (Aerobic Exercise and Computerized Cognitive Training)
Other: Conventional Exercises and Brain health lectures — Participants were exposed to balancing, coordination, stretching, and core exercises. Additionally, they attended brain health lectures to provide a comparative non-interactive cognitive engagement. Both the exercises and lectures were scheduled similar to the intervention group over 12 weeks
  Arms: Control Group

SUMMARY:
Background: Ageing is frequently accompanied by physiological changes that might result in a deterioration in physical and cognitive abilities, which frequently leads to institutionalization or the loss of autonomy. Mild cognitive impairment (MCI) is an intermediate state between normal cognitive aging and early dementia, the optimal period to intervene with preventive strategies and early treatments. Thus, the current study intends to investigate the effects of aerobic and computer-based cognitive training on age-related cognitive decline.

Methods: This is a single-blinded, randomized controlled trial. Elderly patients with mild cognitive impairment (n = 60) will be randomized to 2 arms and treated for 12 weeks: arm 1 (aerobic exercise and computerized cognitive training) and arm 2 (Placebo; will not receive any intervention). Outcome measure used were Montreal Cognitive Assessment (MOCA) test, Barthel Index (BI) and short form survey-12 (SF-12).

Statistical Analysis: To compare the baseline characteristics and outcome variables between the two groups, independent t-tests was employed. A two-way repeated measures ANOVA was utilized to determine the interaction effect of time (baseline, post-treatment, and follow-up) and group (intervention vs. control) on the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Who fulfilled MCI criteria [10]: (1) subjective cognitive concerns; (2) objective cognitive impairment in memory, executive function, attention, and/or language; (3) preserved activities of daily living; and (4) absence of dementia
* Literate
* Had adequate visual, auditory, and fine motor skills.

Exclusion Criteria:

* Major depression (scored > 9 in the Geriatric Depression Scale, GDS-15) [11]
* Schizophrenia
* Substance abuse
* parkinsonism
* conditions affecting gait (eg, severe osteoarthritis, previous stroke),
* participated in any cognitive training program during last 6 months > 2 h/week
* ACSM contraindications to exercise or other factors that make exercise impossible or unsafe
* cognitive enhancers, or anticholinergics

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment test | at the baseline (day 0), at the end of the treatment (after 12 weeks) as well as after 4 weeks of follow up (after 16 weeks)
  A commonly used test to assess different cognitive domains, including short-term memory recall, visuospatial abilities, executive functions, attention, concentration, and working memory. MoCA scores range between 0 and 30 where the highest score is considered to be normal.
Barthel Index | at the baseline (day 0), at the end of the treatment (after 12 weeks) as well as after 4 weeks of follow up (after 16 weeks)
  This index was used to measure an individual's capacity to perform ten activities of daily living, reflecting their functional independence. Total possible scores range from 0 - 20, with lower scores indicating increased disability.
Short form survey-12 | at the baseline (day 0), at the end of the treatment (after 12 weeks) as well as after 4 weeks of follow up (after 16 weeks)
  A generic measure utilized to assess the health-related quality of life, covering both physical and mental health dimensions. The summary scores range from a minimum of 0 to a maximum of 100. Higher the SF-12 scores, indicates the higher (better) quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No